CLINICAL TRIAL: NCT03246841
Title: Investigation of Tumour Spectrum, Penetrance and Clinical Utility of Germline Mutations in New Breast and Ovarian Cancer Susceptibility Genes.
Brief Title: Investigation of Tumour Spectrum of Germline Mutations in Breast and Ovarian Cancer Genes.
Acronym: TUMOSPEC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Institut Curie (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UC-0104/1605 - TUMOSPEC; 2016-A00338-43 (Other: Id-RCB); ONCO04 (Other: UNICANCER)
Record Dates: First submitted 2017-08-04; First posted 2017-08-11 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Hereditary Breast and Ovarian Cancer; Mutation
Keywords: Oncogeneticists; Mutations; Breast Cancer; Ovarian cancer
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Breast Neoplasms; Ovarian Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Analysis of the gene panel (Other): The laboratory will carry out the TUMOSPEC gene panel analysis at the same time as the BRCA1 and BRCA2 analysis and will return a negative (no mutation) or positive (presence of a mutation allowing enrolment of family members) result.
  Interventions: Other: Genetic testing

INTERVENTIONS:
Other: Genetic testing — A panel of 24 genes, chosen in advance by a steering committee, will be tested as the same time as the BRCA1/2 genes, at one of the usual BRCA1/2 analysis laboratories belonging to the same network and participating in the study.

SUMMARY:
TUMOSPEC is a national family study designed to measure the relative and absolute risk of cancer for carriers of deleterious mutations to these "new" breast cancer (BC) susceptibility genes. Index cases will be enrolled consecutively from patients attending an appointment at one of the Unicancer centres, with no other inclusion criteria, and offered a BRCA1/2 analysis as part of their care plan. A panel of 24 TUMOSPEC genes, chosen in advance by a steering committee, will be tested as the same time as the BRCA1/2 genes, at one of the usual BRCA1/2 analysis laboratories belonging to the same network and participating in the study. If a mutation is found, the index cases will be asked to invite their first and second degree family members and their cousins to take part in the study, regardless of whether they have cancer. Saliva samples will be then taken and used for a targeted analysis of the familial abnormality. Each participant will also complete an epidemiological questionnaire in order to gather information about his/her medical history and any exposure to various risk factors. All medical and genotype data will be centralised at the Genetic Epidemiology Research Platform (PIGE, INSERM). The cumulative mutation frequency for all genes is estimated at 10%. Penetrance will be analysed using methods designed to minimise selection bias. The expression spectrum of the mutations will also be described. For genes where the number of mutated families is too low, the data may be contributed to international consortia. The main project will be preceded by a two-year feasibility study, using the same inclusion criteria and logistic circuits. It is this pilot study to which the current funding application relates.

ELIGIBILITY:
Inclusion criteria:

Index case eligibility:

Any person with an indication for a BRCA1/BRCA2 gene analysis and who has been offered TUMOSPEC panel screening.

Age ≥18 years.

Family member eligibility:

Family members will be eligible if the mutation identified in the Index Case is considered deleterious.

Any family member to the first and second decree or a cousin of the Index Case. Family members from both sides of the family will be invited to take part.

Age ≥18 years.

Exclusion Criteria:

People deprived of their civil liberties or who are under judicial protection or guardianship.

Patients unable to answer the questionnaire for social or psychological reasons.

Children of the index cases, of any age.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7274 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Penetrance estimation of the mutations identified in the gene panel | 2 years
  The primary outcome is to obtain unbiased penetrance estimates of the mutations identified in the gene panel (about 20 genes), which will be analysed by the molecular diagnostic laboratories at the same time as the BRCA1 and BRCA2 genes

SECONDARY OUTCOMES:
The results for the whole panel sequencing will be formatted to be used by all laboratories allowing the subsequent centralisation of the data. | 2 years
  This outcome will allow to establish a procedure for centralising homogeneous genomic sequencing data produced by the molecular diagnostics laboratories
Relative risk will be determined by the ratio of calculated cancer incidence in mutated and non-mutated families for this gene. | 2 years
  To determine the deleterious nature of a variant the gene panels will be analysed by the various molecular diagnostics laboratories and we will estimate the relative risk by the ratio of calculated cancer incidence in mutated and non-mutated families for this gene.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CARON, MD, Principal Investigator — Gustave Roussy, Villejuif, France; Andrieu Nadine, PhD, Principal Investigator — Institut Curie, Paris, France; Severine Eon Marchais, PhD, Principal Investigator — PIGE Institut Curie, Paris, France
Locations (2):
- France (2):
  - Gustave Roussy, Paris
  - Institut Curie - PIGE, Paris

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Background] Lesueur F, Eon-Marchais S, Bonnet-Boissinot S, Beauvallet J, Dondon MG, Golmard L, Rouleau E, Garrec C, Martinez M, Toulas C, Nguyen TD, Brayotel F, Crivelli L, Maugard CM, Bubien V, Sevenet N, Gesta P, Chieze-Valero S, Nambot S, Goussot V, Mari V, Popovici C, Prieur F, Morin-Meschin ME, Tinat J, Lortholary A, Dreyfus H, Bidart M, Collonge-Rame MA, Mozelle-Nivoix M, Gladieff L, Giraud S, Boutry-Kryza N, Chiesa J, Denizeau P, Bignon YJ, Uhrhammer N, Cohen-Haguenauer O, Vilquin P, Mailliez A, Coupier I, Rey JM, Lacaze E, Bera O, Colas C, Coulet F, Delnatte C, Houdayer C, Lasset C, Lemonnier J, Longy M, Nogues C, Stoppa-Lyonnet D, Vaur D, Andrieu N, Caron O. TUMOSPEC: A Nation-Wide Study of Hereditary Breast and Ovarian Cancer Families with a Predicted Pathogenic Variant Identified through Multigene Panel Testing. Cancers (Basel). 2021 Jul 21;13(15):3659. doi: 10.3390/cancers13153659. PMID 34359559